CLINICAL TRIAL: NCT05472753
Title: Effect of a Dietary Supplement with Antioxidant and Anti-inflammatory Properties on the Intestinal Microbiota in Patients with Colon Cancer. Randomized, Placebo-controlled Clinical Trial. TERATROPHO Study.
Brief Title: Dietary Supplement on the Intestinal Microbiota in Patients with Colon Cancer
Acronym: TERATROFO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TERATROFO
Record Dates: First submitted 2022-05-04; First posted 2022-07-25 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Colon Cancer
Keywords: intestinal microbiota,; antioxidants; anti-inflammatories
MeSH Terms: conditions — Colonic Neoplasms | interventions — 3,4-dihydroxyphenylethanol; Curcumin; Selenium

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in a 1:1 ratio
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 (25 patients) (Experimental): A product of the company DCOOP, with hydroxytyrosol extract
  Interventions: Dietary Supplement: Experimental Treatment, DCOOP Product, Hydroxytyrosol extract
- Group 2 (25 patients) (Experimental): A product of the company Indukern, with extract of curcumin and selenium
  Interventions: Dietary Supplement: Experimental Treatment,Indukern product, Curcumin and selenium extract
- Group 3 (25 patients) (Placebo Comparator): Placebo
  Interventions: Other: Control Treatment

INTERVENTIONS:
Dietary Supplement: Experimental Treatment, DCOOP Product, Hydroxytyrosol extract — Intervention group will receive a nutritional formula from DCOOP (Spain).
  Arms: Group 1 (25 patients)
Dietary Supplement: Experimental Treatment,Indukern product, Curcumin and selenium extract — Intervention group will receive a nutritional formula from Indukern (Spain).
  Arms: Group 2 (25 patients)
Other: Control Treatment — Control group will receive a placebo (product loading substance)
  Arms: Group 3 (25 patients)

SUMMARY:
Effect of a dietary supplement with antioxidant and anti-inflamatory properties on the intestinal microbiota in patients with colon cancer. Ramdonized placebo controlled clinical trial. Teratrophic study

DETAILED DESCRIPTION:
Introduction:

The alteration in the microbiota plays a fundamental role in the promotion and progression of colon cancer due to various pathways such as inflammation and oxidative stress. The use of substances with anti-inflammatory and antioxidant effect could be useful for the treatment of this disease.

Methodology:

Prospective randomized clinical trial, with three parallel groups and double blind. Patients with stage II or III colon neoplasia who are going to receive post-surgical chemotherapy will be included. Patients will be randomized to one of the following groups: group 1 (25 patients): product with hydroxytyrosol extract; group 2 (25 patients): product with curcumin and selenium extract. Group 3 (25 patients): placebo. Before starting chemotherapy, stool and blood samples will be taken, and gastrointestinal symptoms, quality of life, symptoms of anxiety-depression and evaluation of nutritional status will be assessed. When starting chemotherapy, they will start with a daily intake of the assigned dietary supplement. At 3 months ± 2 weeks after starting chemotherapy (at least 2 weeks must have passed since the last chemotherapy of the fourth cycle), the same assessment will be made as in the initial visit, in addition to recording adherence to the intervention dietary supplement and new health problems that have appeared since the previous visit.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stage II or III colo neoplasia
* Indication of adjuvant chemotherapy according to the Protocols for the diagnosis and treatment of cancer of the Intercenter Clinical Management Unit
* Sign the informed consent

Exclusion Criteria:

* Systemic autoimmune diseases (systemic lupus erythematosus, antiphospholipid syndrome, Sjögren's syndrome, progressive systemic sclerosis -scleroderma-, idiopathic inflammatory myopathies -myositis-, vasculitis, Behçet's disease, relapsing polychondritis, etc.)
* Mellitus diabetes type 1
* Previous gastrointestinal resections, except for appendectomy or surgery required to treat colon neoplasia
* Chronic intestinal pathologies (inflammatory bowel disease, celiac disease, lymphangiectasias)
* Continued consumption of probiotics, with the exception of dairy products or other natural fermented foods
* Chronic and continued use of NSAIDs or corticosteroids
* Allergy to any component of the product under investigation
* Pregnancy
* Mean consumption of > 3 UBE of alcohol per day
* Previous or concomitant neoplasia, unless curative treatment was received and ≥5 years have passed free of disease
* ECOG scale greater than or equal to 3 at the start of the clinical trial
* Grade 3-4 neuropathy that limits the use of oxaliplatin.
* History of familial adenomatous polyposis mediated by the APC gene or by Lynch syndrome (mutations MLH1, MSH2, PMS2, MSH6).
* Patients with partial or complete deficiency of the enzyme dihydropyrimidine dehydrogenase (DPD), which causes poor metabolism and the use of fluoropyrimidines is contraindicated.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2022-11-16 (Actual); Primary Completion 2024-02-27 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Change in the alpha diversity index (Shannon) | From baseline to 3 months about 2 weeks after starting chemotherapy
  This diversity index is a quantitative indicator of the number of different bacteria that are present in a stool sample, taking into account the uniformity in the distribution of these bacteria in these species. Diversity index value increases both when the number of species increases and when evenness increases. The Shannon index is a well-known diversity index used in microecological studies. The higher the Shannon index value, the higher the community diversity. It is calculated as: H = -Σpi * ln(pi), where "H" is the Shannon Diversity Index. "Σ" is a Greek symbol that means "sum". "ln" is natural log. "pi" is the proportion of the entire community made up of species i. The minimum value the Shannon diversity index can take is 0. Such a number would tell us that there is no diversity - only one species is found in that habitat. There is no upper limit to the index.

SECONDARY OUTCOMES:
Change in weight | From baseline to 3 months about 2 weeks after starting chemotherapy
  Weight in kg
Change in height | From baseline to 3 months about 2 weeks after starting chemotherapy
  Height in m
BMI (body mass index) changes | From baseline to 3 months about 2 weeks after starting chemotherapy
  Measured by body composition analysis
Mediterranean diet adherence questionnaire | From baseline to 3 months about 2 weeks after starting chemotherapy
  to evaluate adherence to a Mediterranean diet pattern. It consists of 14 items in which different components of the Mediterranean diet are evaluated (number of pieces of fruit consumed per day, number of portions of legumes consumed per week...). Each item is scored as 0 or 1. A total score of <9 indicates poor adherence, while a score of ≥9 indicates good adherence.
Maximum and mean value of 3 measurements in dominant hand dynamometry | From baseline to 3 months about 2 weeks after starting chemotherapy
  Measured in kg
Maximum and mean value of 3 measurements in non dominant hand dynamometrydynamometry | From baseline to 3 months about 2 weeks after starting chemotherapy
  Measured in kg
Mean dominant arm circumference | From baseline to 3 months about 2 weeks after starting chemotherapy
  Measured in cm
Calf circumference in the dominant leg | From baseline to 3 months about 2 weeks after starting chemotherapy
  Measured in cm
Anteroposterior diameter of the rectus femoris of the quadriceps in the dominant thigh | From baseline to 3 months about 2 weeks after starting chemotherapy
  Measured in cm
Transverse diameter of the rectus femoris of the quadriceps in the dominant thigh | From baseline to 3 months about 2 weeks after starting chemotherapy
  Measured in cm
Cross-sectional area of the rectus femoris quadriceps in the dominant thigh | From baseline to 3 months about 2 weeks after starting chemotherapy
  Measured in in cm²
Transverse perimeter of the quadriceps rectus muscle in the dominant thigh | From baseline to 3 months about 2 weeks after starting chemotherapy
  Measured in cm
Mean value of 3 measurements of the anteroposterior diameter of abdominal subcutaneous adipose tissue | From baseline to 3 months about 2 weeks after starting chemotherapy
  Measured in cm
Mean value of 3 measurements of the anteroposterior diameter of abdominal visceral adipose tissue | From baseline to 3 months about 2 weeks after starting chemotherapy
  Measured in cm
Fat mass in bioimpedanciometry | From baseline to 3 months about 2 weeks after starting chemotherapy
  Measured in kg
Lean mass in bioimpedanciometry | From baseline to 3 months about 2 weeks after starting chemotherapy
  Measured in kg
Extracellular water in bioimpedanciometry | From baseline to 3 months about 2 weeks after starting chemotherapy
  Measured in kg
Phase angle 50 kHz in bioimpedance measurement | From baseline to 3 months about 2 weeks after starting chemotherapy
  Measured in º
Total cell mass in bioimpedance measurement | From baseline to 3 months about 2 weeks after starting chemotherapy
  Measured in kg
Appendicular muscle mass in bioimpedanciometry | From baseline to 3 months about 2 weeks after starting chemotherapy
  Measured in kg
Percentage of weight lost in the last 6 months | From baseline to 3 months about 2 weeks after starting chemotherapy
  Measured in %.
Percentage of weight lost in the last 12 months | From baseline to 3 months about 2 weeks after starting chemotherapy
  Measured in %.
Hemoglobin in blood | From baseline to 3 months about 2 weeks after starting chemotherapy
  Measured in g/dl
Mean corpuscular volume in blood | From baseline to 3 months about 2 weeks after starting chemotherapy
  Measured in in fL
Leukocytes in blood | From baseline to 3 months about 2 weeks after starting chemotherapy
  Measured in in x10^9/l
Lymphocytes in blood | From baseline to 3 months about 2 weeks after starting chemotherapy
  Measured in in x10^9/l
Platelets in blood | From baseline to 3 months about 2 weeks after starting chemotherapy
  Measured in in x10^9/l
Creatinine in blood | From baseline to 3 months about 2 weeks after starting chemotherapy
  Measured in in g/dl
Glucose in blood | From baseline to 3 months about 2 weeks after starting chemotherapy
  Measured in in mg/dl
Sodium in blood | From baseline to 3 months about 2 weeks after starting chemotherapy
  Measured in mEq/l
Potassium in blood | From baseline to 3 months about 2 weeks after starting chemotherapy
  Measured in mEq/l
Chlorine in blood | From baseline to 3 months about 2 weeks after starting chemotherapy
  Measured in mEq/l
Calcium in blood | From baseline to 3 months about 2 weeks after starting chemotherapy
  Measured in in mg/dl
Phosphorus in blood | From baseline to 3 months about 2 weeks after starting chemotherapy
  Measured in in mg/dl
Magnesium in blood | From baseline to 3 months about 2 weeks after starting chemotherapy
  Measured in in mg/dl
Iron in blood | From baseline to 3 months about 2 weeks after starting chemotherapy
  Measured in in mcg/dl
Blood cholesterol | From baseline to 3 months about 2 weeks after starting chemotherapy
  Measured in in mg/dl
HDL cholesterol in the blood | From baseline to 3 months about 2 weeks after starting chemotherapy
  Measured in in mg/dl
LDL cholesterol in the blood | From baseline to 3 months about 2 weeks after starting chemotherapy
  Measured in in mg/dl
Blood triglycerides | From baseline to 3 months about 2 weeks after starting chemotherapy
  Measured in in mg/dl
ALT in blood | From baseline to 3 months about 2 weeks after starting chemotherapy
  Measured in U/L
GGT in blood | From baseline to 3 months about 2 weeks after starting chemotherapy
  Measured in U/L
Alkaline phosphatase in blood | From baseline to 3 months about 2 weeks after starting chemotherapy
  Measured in U/L
Bilirubin in blood | From baseline to 3 months about 2 weeks after starting chemotherapy
  Measured in mg/dl
Total protein in blood | From baseline to 3 months about 2 weeks after starting chemotherapy
  Measured in g/dl
Albumin in blood | From baseline to 3 months about 2 weeks after starting chemotherapy
  Measured in g/dl
Ferritin in blood | From baseline to 3 months about 2 weeks after starting chemotherapy
  Measured in ng/ml
25OH vitamin D in blood | From baseline to 3 months about 2 weeks after starting chemotherapy
  Measured in ng/ml
Prealbumin in blood | From baseline to 3 months about 2 weeks after starting chemotherapy
  Measured in mg/dl
C-reactive protein in blood | From baseline to 3 months about 2 weeks after starting chemotherapy
  Measured in mg/dl
Normalized prothrombin time | From baseline to 3 months about 2 weeks after starting chemotherapy
  Measured in in INR
Degree in "ECOG Performance Status Scale" | From baseline to 3 months about 2 weeks after starting chemotherapy
  This scale was developed by the Eastern Cooperative Oncology Group (ECOG), currently the ECOG-ACRIN Cancer Research Group. It was published in 1982. The scale describes the level of functioning of a patient in terms of her ability to take care of herself, perform daily physical activity and physical capacity (walk, work…). It was devised to use standard criteria between different centers to measure how the disease affects a patient's daily living abilities. The scale has a score from 0 to 5 in whole numbers. Lower score indicates better functional capacity. Score 0 refers to fully active patients, capable of carrying out all activities as before the onset of the disease. A score of 5 indicates the death of the patient.
Assess the effect of supplementation on quality of life: "EORTC QLQ-30" test. | From baseline to 3 months about 2 weeks after starting chemotherapy
  The "EORTC quality of life questionnaire (QLQ)" is an integrated system to assess the quality of life of cancer patients participating in international clinical trials. The main questionnaire is the "QLQ-C30". Version 3.0 is currently the standard version. The QLQ-C30 is made up of multiple-item and single-item scales. Five functionality scales, three symptom scales, a global health status/quality of life scale, and six individual items are included. Each of the multiple item scales includes a different set of items; no item appears on more than one scale. All single-item scales and measures range in score from 0 to 100. A high scale score represents a higher level of response. Thus, a high score for a functionality scale represents a high/healthy level of functionality, a high score for global health status/quality of life represents a high quality of life, but a high score for a scale or isolated items of symptoms represents a high level of symptoms/problems.
Assess the effect of supplementation on quality of life: "EORTC QLQ-CR29" test. | From baseline to 3 months about 2 weeks after starting chemotherapy
  It is a supplemental questionnaire module to be used together with the QLQ-C30. The QLQ-CR29 incorporates 4 multi-item and 19 single-item scales. A variety of common symptoms and problems are assessed in colorectal cancer patients. The scoring approach is identical in principle to that of the scales or isolated items of functionality and symptoms of the QLQ-C30. All scales and single-item measures have a score range of 0 to 100. A high score on the functionality scale and the isolated items of functionality represents a high level of functionality, while a high score for the scales and isolated items represents a high level of functionality. of symptoms represents a high level of symptomatology or problems.
Assess the effect of supplementation on symptoms of depression-anxiety | From baseline to 3 months about 2 weeks after starting chemotherapy
  Hospital Anxiety and Depression Scale (HADS). Its objective is to detect depressive and anxious disorders in non-psychiatric hospital services, avoiding overlapping with symptoms due to physical illness, without taking into account the physical aspects that may accompany anxiety/depression, focusing only on emotional ones. It is a self-administered scale with 14 items divided into 2 subscales (anxiety and depression) whose maximum score is 21 points for each of them. Based on the score obtained, patients can be classified as normal (<7), doubtful (between 8 and 10) and potential clinical case (≥11). The score is referred to the last week.
Assess gastrointestinal tolerance to supplementation and chemotherapy | From baseline to 3 months about 2 weeks after starting chemotherapy
  Gastrointestinal symptoms questionnaire: an own questionnaire created for this study will be carried out in which the presence of nausea, vomiting, diarrhoea, constipation, acid reflux, early satiety, abdominal distension and abdominal pain will be evaluated. Each variable is evaluated on a scale with 4 possible responses: absent, mild, moderate, severe.
Change in serum C-reactive protein | From baseline to 3 months about 2 weeks after starting chemotherapy
  Measured in mg/l
Change in serum Il-6 | From baseline to 3 months about 2 weeks after starting chemotherapy
  Measured in pg/ml
Change in serum TNF-alpha | From baseline to 3 months about 2 weeks after starting chemotherapy
  Measured in pg/ml
Change in stool calprotectin | From baseline to 3 months about 2 weeks after starting chemotherapy
  Measured in mcg/g

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Olveira Fuster, MD, PhD., Principal Investigator — Hospital Regional Universitario de Málaga, FIMABIS
Locations (1):
- Hospital Regional Universitario de Málaga, Málaga, Málaga, Spain